CLINICAL TRIAL: NCT03681379
Title: Pharmacokinetics of Levosimendan, OR1855 and OR1896 in Neonates and Children With or Without Extracorporeal Membrane Oxygenation
Brief Title: Pharmacokinetics of Levosimendan in Pediatric Intensive Care Units
Acronym: PALMAréa
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC16_0114
Record Dates: First submitted 2018-09-18; First posted 2018-09-24 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Acute Heart Failure
Keywords: Levosimendan; pharmacokinetics; children; acute heart failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients with acute circulatory insufficiency are equipped with a central venous line or catheterization for hemodynamic monitoring and biological assessment in context of routine care. There will be no specific interventions to the study participants like additional venipuncture for this study. The volume required for the analyzes (0.5 ml, 13 times over a period of 8 days) are issue from hemodynamic monitoring and biological assessment in context of routine care . This volume is compatible with the current french regulation on non interventional research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To describe pharmacokinetics of levosimendan in neonates and children supported or not with extracorporeal circulation devices (ECMO, CRRT)

DETAILED DESCRIPTION:
Levosimendan is a calcium sensitiver wih inotropic effects. It's use in the context of acute or chronic heart failure in children has yet to be defined. Due to physical proprieties of levosimendan and metabolites, we hypothesized that concomitant use of extracorporeal devices such as ECMO will cause major pharmacokinetic variations. Furthermore, pharmacokinetics of levosimendan in children with multiple organ failure has to be specify.

ELIGIBILITY:
Inclusion Criteria:

* All children admitted in pediatric intensive care units with planned infusion of 0.2 mcg/kg/min of levosimendan over 24h in context of routine care
* Arterial line or central venous catheter inserted for blood sampling procedures in context of routine care.

Exclusion Criteria:

* Absence of clear parental status or information

Ages: 0 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children admitted in pediatric intensive care units for acute heart failure
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2018-09-23 (Actual); Primary Completion 2019-10-11 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
First parameter of the pharmacokinetics of levosimendan, OR1855, OR1896 (Area under the plasma concentration versus time curve (AUC) ) | At the end of the study, after 2 years.
  Area under the plasma concentration versus time curve (AUC) of levosimendan, OR 1855 and OR 1896. Samples will be collected over a period in of 192h in context of routine care
second parameter of the pharmacokinetics of levosimendan, OR1855, OR1896 (distribution volume) | At the end of the study, after 2 years.
  distribution volume of levosimendan, OR 1855 and OR 1896. Samples will be collected over a period in of 192h in context of routine care
third parameter of the pharmacokinetics of levosimendan, OR1855, OR1896 (half-life time) | At the end of the study, after 2 years.
  half-life time of levosimendan, OR 1855 and OR 1896. Samples will be collected over a period in of 192h in context of routine care
fourth parameter of the pharmacokinetics of levosimendan, OR1855, OR1896 (Peak Plasma Concentration (Cmax)) | At the end of the study, after 2 years.
  Peak Plasma Concentration (Cmax) of levosimendan, OR 1855 and OR 1896. Samples will be collected over a period in of 192h in context of routine care

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kivikko M, Antila S, Eha J, Lehtonen L, Pentikainen PJ. Pharmacokinetics of levosimendan and its metabolites during and after a 24-hour continuous infusion in patients with severe heart failure. Int J Clin Pharmacol Ther. 2002 Oct;40(10):465-71. doi: 10.5414/cpp40465. PMID 12395979
- [Derived] Bourgoin P, Lecomte J, Oualha M, Berthomieu L, Pereira T, Davril E, Lamoureux F, Joram N, Chenouard A, Duflot T. Population Pharmacokinetics of Levosimendan and its Metabolites in Critically Ill Neonates and Children Supported or Not by Extracorporeal Membrane Oxygenation. Clin Pharmacokinet. 2023 Feb;62(2):335-348. doi: 10.1007/s40262-022-01199-y. Epub 2023 Jan 11. PMID 36631687